CLINICAL TRIAL: NCT01344070
Title: Generic Formulations of Commonly-Used, Immediate-Release, Solid, Oral, Drugs in Saudi Arabia: Interchangeability & Post-Marketing Quality
Brief Title: Generic Formulations of Commonly-used Oral Drugs in Saudi Arabia:Interchangeability & Post-marketing Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Collaborators: Saudi National Comprehensive Plan for Science & Technology (Unknown)
Responsible Party: Principal Investigator, Muhammad Maher Hammami, Chairman, Department of Clinical Studies & Empirical Ethics, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: RAC 2101100; project 10-BIO961-20 (Other Grant/Funding Number: Saudi National Comprehensive Plan for Science & Technology)
Record Dates: First submitted 2011-04-03; First posted 2011-04-28 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Generic Drug Quality; Generic Formulation Interchangeability
Keywords: innovator formulations; generic formulations; bioequivalence; interchangeability; inter-patch variation; quality of generic drug formulations on the market; Interchangeability between marketed generic formulations; prevalence of large intrasubject variability despite average bioequivalence; Causes of large intrasubject variability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Reference formulation of each drug (Active Comparator): Innovator formulation
  Interventions: Drug: one of the 15 drugs listed below
- generic formulation a (Active Comparator): one of the several generic formulations in the market, randomly selected for each drug
  Interventions: Drug: one of the 15 drugs listed below
- generic formulation b (Active Comparator): second of the several generic formulations in the market, randomly selected for each drug
  Interventions: Drug: one of the 15 drugs listed below
- generic formulation c (Active Comparator): third of the several generic formulations in the market, randomly selected for each drug
  Interventions: Drug: one of the 15 drugs listed below

INTERVENTIONS:
Drug: one of the 15 drugs listed below — single, oral, immediate-release, non-combinational innovator formulation
  Arms: Reference formulation of each drug
Drug: one of the 15 drugs listed below — single, oral, immediate-release, non-combinational generic formulation a
  Arms: generic formulation a
Drug: one of the 15 drugs listed below — single, oral, immediate-release, non-combinational generic formulation b
  Arms: generic formulation b
Drug: one of the 15 drugs listed below — single, oral, immediate-release, non-combinational generic formulation c
  Arms: generic formulation c

SUMMARY:
Generic formulations of prescription drugs can, through their relatively lower cost, improve healthcare as long as they maintain their registration-quality and public trust. On the other hand, the market availability of several generic formulations raises a concern regarding their interchangeability, despite being proven to be individually therapeutically interchangeable with their corresponding innovator formulation.

The investigators propose to assess the quality and therapeutic interchangeability of generic formulations in the drug market of Saudi Arabia, using fifteen, commonly-used, oral, solid, immediate-release, and non-combinational drugs.

DETAILED DESCRIPTION:
Generic formulations of prescription drugs can, through their relatively lower cost, improve healthcare as long as they maintain their registration-quality and public trust. On the other hand, the market availability of several generic formulations raises a concern regarding their interchangeability, despite being proven to be individually therapeutically interchangeable with their corresponding innovator formulation.

The investigators propose to assess the quality and therapeutic interchangeability of generic formulations in the drug market of Saudi Arabia, using fifteen, commonly-used, oral, solid, immediate-release, and non-combinational drugs.

The following drugs have been identified from the Saudi National Formulary (September 2006) as having, among oral, immediate-release, non-combinational drugs, the highest number of formulations (they have each 15 to 47): ciprofloxacin, ranitidine, amoxicillin, paracetamol, atenolol, cephalexin, ibuprofen, diclofenac, metformin, omeprazole, metronidazole, enalapril, clarithromycin, amlodipine, and fluconazole. In the first set of studies and for each drug, a four-treatment, four-period, four-sequence, crossover bioequivalence study will be conducted on the innovator and three randomly-selected generic formulations. Each study will be designed to have a power of 0.9 to detect bioequivalence, and sampling and wash-out periods of at least 5 and 7 half lives, respectively. Individuals who are identified in the first set of studies as having the large intra-subject variation (bioequivalence parameters ratios of less the 80% or more than 120% for AUC) will be subjected to a second set of studies, in which 2 batches of the reference formulation (including the batch used in the first set of studies) and the generic formulation will be compared in a two-treatment, four-period, two-sequence, replicate design crossover bioequivalence study. Drug levels will be determined by an HPLC or LC-MS-MS method, locally-validated according to international guidelines. After log transformation, AUC and Cmax (non-compartmental model) of the formulations will be compared pair-wise by ANOVA. Pair-wise bioequivalence will be tested by 90% (and 95%) confidence interval of ratios and Schuirmann's two one sided t-tests for the 70-143, 80-125%, and 90-112% ranges. The following will be determined: 1) the prevalence of generic formulations that are not bioequivalent to their innovator formulation, 2) the prevalence of the phenomena that two generics of the same innovator formulation are not bioequivalent to each other, 3) the percentage of individuals with large intra-subject variation despite the presence of average bioequivalence between the two formulations, and 4) how much of the large intra-subject variation in 3 above is true or related, in part, to product failure, random error, or subject-by-formulation interaction; and how it compares to intra-subject variability when two batches of the innovator formulation are compared.

ELIGIBILITY:
Inclusion Criteria:

* No evidence of clinically important deviation from normal health as indicated by a recent physical examination, medical history, and clinical laboratory tests (complete blood count, renal and hepatic profiles, and routine urinalysis.
* Body Mass Index (BMI) should be less than 35 kg/m2.
* Acceptance to abstain from taking any medication (including over-the-counter [OTC] drugs) for at least 2 weeks prior to, and during the study; and from smoking and taking alcohol or caffeine or related xanthenes-containing beverages or food for 48 hours before taking the study drug and throughout each of the two blood sampling periods.

Exclusion Criteria:

* any contraindication to use the drug.
* any history of hypersensitivity to the drug to be tested or related compounds.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2011-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
bioequivalence | ciprofloxacin 24hrs,ranitidine 14hrs,amoxicillin 10hrs,paracetamol 14hrs,atenolol 36hrs,cephalexin 6hrs,ibuprofen 10hrs,diclofenac 14hrs,metformin 32hrs,omperazole 12hrs,metronidazole 48hrs,enalapril 8hrs,clarithromycin 24hrs,amlodipine 240hrs
  Bioequivalence between marketed generic formulations and their corresponding innovator formulations and between 2 marketed generic formulations. Bioequivalence will be assessed by the ratio of the area under the curve (AUC) (drug level vs time)and maximum levels (cmax) of two formulations and analyzed by the 90% confidence interval method. The time is 3-5 plasma half-life of each drug.
Intra-subject variation despite average bioequivalence | ciprofloxacin 24hrs,ranitidine 14hrs,amoxicillin 10hrs,paracetamol 14hrs,atenolol 36hrs,cephalexin 6hrs,ibuprofen 10hrs,diclofenac 14hrs,metformin 32hrs,omperazole 12hrs,metronidazole 48hrs,enalapril 8hrs,clarithromycin 24hrs,amlodipine 240hrs
  Large intra-subject variation (a ratio of the test to reference formulation of AUC that is less than 80% or more than 120%) between innovator and generic formulation, despite showing average bioequivalence between the two formulations

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad M Hammami, MD, PhD, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Hammami MM, De Padua SJS, Hussein R, Al Gaai E, Khodr NA, Al-Swayeh R, Alvi SN, Binhashim N. Generic-reference and generic-generic bioequivalence of forty-two, randomly-selected, on-market generic products of fourteen immediate-release oral drugs. BMC Pharmacol Toxicol. 2017 Dec 8;18(1):78. doi: 10.1186/s40360-017-0182-1. PMID 29216899